CLINICAL TRIAL: NCT02566746
Title: Contribution of Percutaneous Endoscopic Caecostomie in the Management of Severe Constipation Refractory to Medical Treatment
Acronym: ConstiCAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC15_0041
Record Dates: First submitted 2015-10-01; First posted 2015-10-02 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chait Trapdoor caecostomie catheter (Experimental): Patients randomized in this arm will undergo percutaneous endoscopic caecostomy with Chait Trapdoor caecostomie catheter
  Interventions: Device: Chait Trapdoor caecostomie catheter
- Continuation of optimal medical therapy (Active Comparator): Patients randomized in this arm will continue this medical treatment of constipation with laxative and / or suppositories and / or enemas retrograde during 12 months.
  At 12 months : patients will undergo percutaneous endoscopic caecostomy with Chait Trapdoor caecostomie catheter during 12 months.
  Interventions: Device: Chait Trapdoor caecostomie catheter; Drug: continuation of optimal medical therapy

INTERVENTIONS:
Device: Chait Trapdoor caecostomie catheter — implantation of the Chait Trapdoor caecostomie catheter
Drug: continuation of optimal medical therapy — continuation of treatment with laxative and / or suppositories and / or enemas retrograde At 12 months : implantation of the Chait Trapdoor caecostomie catheter
  Other Names: Chait Trapdoor caecostomie catheter
  Arms: Continuation of optimal medical therapy

SUMMARY:
The investigators' study aims to compare the results of percutaneous endoscopic caecostomie (CPE) to optimal medical therapy in the treatment of patients with constipation refractory to medical treatment. The primary endpoint will be the quality of life assessed by the Gastrointestinal Quality Of Life Index (GIQLI) at one year. The secondary endpoints are digestive symptoms, Kess's constipation scores and Cleveland's incontinence score, tolerance of the Chait TrapdoorTM caecostomy catheter (CTCC) and the collection of possible complications. The patients included must meet the classification criteria of Rome III, have an elongated colonic transit time, have had a complete colonoscopy and be refractory to medical treatment including at least one stimulant laxative or suppositories or enemas retrograde.

ELIGIBILITY:
Inclusion Criteria:

* Patient betwen 18 and 75 years old
* Chronic constipation defined by the Rome III classification
* Transit time with pellets made within 24 months preceding the inclusion visit indicating a transit time of at least 120 hours and/or with a Neurogenic bowel dysfunction ≥ 14 for patients with spina bifida and / or spinal cord injuries.
* Colonoscopy made within the 5 years preceding the inclusion visit indicating the absence of colorectal organic obstacle
* Anorectal manometry performed within 24 months preceding the inclusion visit performed to substantiate the information on the type of constipation
* GIQLI score <121 and Kess Questionnaire score> 7, despite medical treatment of constipation including taking a laxative (stimulant laxative orally and / or suppository and / or retrograde enema) more than one times per week for at least two months.
* Affiliation to a social security
* - Chronic constipation defined by the Rome III classification
* Transit time with pellets made within 24 months preceding the inclusion visit indicating an increase of at least 120 hours compared to normal
* Colonoscopy made within the 24 months preceding the inclusion visit indicating the absence of colorectal organic obstacle
* Anorectal manometry performed in the 24 months preceding the inclusion visit performed to substantiate the information on the type of constipation
* Score GIQLI love <121 and Kess Questionnaire score> 7, despite medical treatment of constipation including taking a laxative (stimulant laxative orally and / or suppository and / or retrograde enema) more than one times per week for at least two months.
* Affiliation to a social security scheme
* Informed consent signed

Exclusion Criteria:

* Severe obesity (BMI> 40)
* History of surgical resection of colon
* Hypothyroidism, electrolyte disorders, insulin-dependent diabetes
* Acute decompensation of depressive syndrome
* Immunosuppressive therapy
* Disorders of hemostasis (TP <70%, APTT> 1.5, thrombocytopenia <70,000 / mm3)
* Pregnant woman (positive serum beta-hCG) or breastfeeding
* Adults under guardianship, curatorship or under court protection
* Participation in another research protocol on the treatment of constipation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Quality of life (Gastrointestinal Quality Of Life Index) | 1 year
  assessed by the Gastrointestinal Quality Of Life Index (GIQLI)

SECONDARY OUTCOMES:
Quality of life (Gastrointestinal Quality Of Life Index) | 21 months
  Evolution of quality of life assessed by the Gastrointestinal Quality Of Life Index (GIQLI)
Evolution of the Quality of life (SF-36 score) | 2 years
  Evolution of the SF-36 score
Constipation score (Kess score) | 2 years
  Evolution of the Kess score
Incontinence score (Cleveland score) | 2 years
  Evolution of the Cleveland score
Neurogenic bowel dysfunction score | 2 years
  Evolution of the Neurogenic bowel dysfunction score for patients with spina bifida and / or spinal cord injuries
Tolerance to the CTCC (Visual Analogue Scale) | 2 years
  Evolution of the tolerance to the CHAIT Trapdoor caecostomy catheter on a skin and abdominal level with Visual Analogue Scale
Constipation treatments | 2 years
  Type of constipation treatments taken by the patient during the study and analysis of compliance
Complications | 2 years
  Reports of immediate or delayed complications

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU de Nantes, Nantes
  - CMRRF de Kerpape, Ploemeur
  - CHU de Rouen, Rouen

REFERENCES:
- [Derived] Lefevre C, Le Roy C, Bessard A, Le Berre-Scoul C, Marchix J, Coron E, Le Rhun M, Brochard C, Perrouin-Verbe B, Neunlist M. Region-specific remodeling of the enteric nervous system and enteroendocrine cells in the colon of spinal cord injury patients. Sci Rep. 2023 Oct 6;13(1):16902. doi: 10.1038/s41598-023-44057-y. PMID 37803037